CLINICAL TRIAL: NCT04624048
Title: "Influence of Physical Exercise on the Severity of Severe Acute Respiratory Syndrome Coronavirus 2 Infection, COVID-19"
Brief Title: Exercise Influence on COVID-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, CARLOS MARTIN SANCHEZ, Doctor, University of Salamanca
Other Study IDs: 08112020
Record Dates: First submitted 2020-11-08; First posted 2020-11-10 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Infection Viral; Exercise; Coronavirus; Habits
Keywords: Exercise; Universities; Coronavirus; Habits
MeSH Terms: conditions — Virus Diseases; Motor Activity; Coronavirus Infections; Habits

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- University population: Survey to analyze the impact of COVID-19.
  Interventions: Diagnostic Test: COVID-19 survey

INTERVENTIONS:
Diagnostic Test: COVID-19 survey — Participants should complete a survey to analyze the impact of COVID-19 on University population.

SUMMARY:
An observational study is carried out in the university population of the University of Salamanca to know the impact of the COVID-19 pandemic and the influence of physical exercise on the severity of symptoms.

DETAILED DESCRIPTION:
* Investigate the relationship between the regular practice of moderate physical exercise and the severity of the COVID-19 disease in the university community of the University of Salamanca.
* Prepare an epidemiological study of the impact of the pandemic at the University of Salamanca.
* Analyze the influence of the pandemic on the sports habits of the university community.
* The study population will be the entire university community (teaching and research staff, administration and services staff, and students) who will be contacted via email.

ELIGIBILITY:
Inclusion Criteria:

* University of Salamanca population
* Complete the survey

Exclusion Criteria:

* Survey not filled out completely

Ages: 17 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: University of Salamanca population, which includes:
  * Teaching and research staff
  * Administration and services staff
  * Students
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2020-12-04 (Estimated); Primary Completion 2021-01-04 (Estimated); Study Completion 2021-04-04 (Estimated)

PRIMARY OUTCOMES:
Impact of COVID-19 | Through study completion, an average of 3 months
  Number of positives

SECONDARY OUTCOMES:
Influence of exercise in COVID-19 infection | Through study completion, an average of 3 months
  Quantity of physical exercise
Change in the practice of physical exercise after home confinement | Through study completion, an average of 3 months
  Change at exercise habits on University population

CONTACTS AND LOCATIONS:
Overall Officials: CARLOS MARTIN-SANCHEZ, DOCTOR, Principal Investigator — University of Salamanca

IPD SHARING:
Plan to Share IPD: Undecided
It will be decided when the recruitment period ends.

REFERENCES:
- [Background] McAuley PA, Keteyian SJ, Brawner CA, Dardari ZA, Al Rifai M, Ehrman JK, Al-Mallah MH, Whelton SP, Blaha MJ. Exercise Capacity and the Obesity Paradox in Heart Failure: The FIT (Henry Ford Exercise Testing) Project. Mayo Clin Proc. 2018 Jun;93(6):701-708. doi: 10.1016/j.mayocp.2018.01.026. Epub 2018 May 3. PMID 29731178